CLINICAL TRIAL: NCT05535348
Title: Evaluation of a Resiliency Program for Fathers of Children and Youth With Special Health Care Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Kuhlthau, Professor, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022P000562
Record Dates: First submitted 2022-06-25; First posted 2022-09-10 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Stress; Family; Fathers

STUDY DESIGN:
Intervention Model Description: We ran two groups of a resiliency intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Pilot (Experimental): An adapted version of the Relaxation Response Resiliency Program (3RP) for fathers of CYSHCN. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Interventions: Behavioral: Relaxation Response Resiliency Program for Father of CYSHCN

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Program for Father of CYSHCN — Virtually delivered psycho-educational resiliency training program for fathers of CYSHCN

SUMMARY:
Based on findings from our prior trials with parents of children with learning and attentional disabilities and parents of children with autism spectrum disorder (Kuhlthau et al., 2020; Park et al., 2020; IRB approved: #:2016P001622 and 2016P002037 respectively), the investigators propose to pilot test and refine the adapted resiliency intervention (SMART-3RP) among fathers of children with special health care needs.

DETAILED DESCRIPTION:
This is an open pilot study. Based on Phase I findings (IRB #2021P002838), the investigators propose to enroll up to 12 fathers (in 2 groups) of children and youth with special health care needs (CYSHCN) in the adapted SMART-3RP intervention. The SMART-3RP is an 8-session mind-body resiliency intervention that will be conducted virtually. Participants will complete the study survey at baseline and immediately following the intervention. As this is a pilot, participants will also be asked to provide weekly feedback on program sessions and participate in an exit interview following the intervention. The intervention may be iteratively modified as the investigators receive feedback from participants.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported identify as father or male guardian of at least one child with special health care needs (e.g., autism spectrum disorder, cerebral palsy, dyslexia)
* Age 18 or older
* Ability to participate in group, virtual sessions including access to computer, tablet, or smartphone and internet.

Exclusion Criteria:

* unable to speak or read English
* unwilling or unable to participate in the study
* considered medically or otherwise unable to participate by the study PI.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported identify as father or male guardian of at least one child with special health care needs (e.g., autism spectrum disorder, cerebral palsy, dyslexia)
Enrollment: 14 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Feedback regarding adapted intervention acceptability by session | 6 months
  Likert ratings on post-session feedback surveys (0 to 5 with 5 more acceptable), qualitative responses from exit interviews

SECONDARY OUTCOMES:
Feasibility (attendance at 6/8 sessions) | 8 weeks
  Feasibility will be assessed using attendance (i.e. 6/8 sessions).
Feasibility (data collection number completing study surveys) | 3 months
  Feasibility will be assessed using number of dads completing study surveys
Acceptability helpfulness ratings of sessions and aspects of program | 3 months
  Acceptability will be assessed using a Participant Feedback questionnaire: questionnaire includes ratings of session helpfulness (1 to 5 with 1 being very helpful and 1 being not at all helpful), likert ratings of program aspects (number, length, etc of sessions), and open-ended qualitative feedback questions.

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Kuhlthau, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuhlthau KA, Luberto CM, Traeger L, Millstein RA, Perez GK, Lindly OJ, Chad-Friedman E, Proszynski J, Park ER. A Virtual Resiliency Intervention for Parents of Children with Autism: A Randomized Pilot Trial. J Autism Dev Disord. 2020 Jul;50(7):2513-2526. doi: 10.1007/s10803-019-03976-4. PMID 30900195
- [Result] Luberto CM, Perez GK, Finkelstein-Fox L, Millstein RA, Fell L, Chad-Friedman E, Park ER, Kuhlthau KA. Acceptability of a Virtual Mind-Body Intervention for Parents of Children With Autism or Learning Disabilities. Glob Adv Health Med. 2021 Dec 9;10:21649561211047804. doi: 10.1177/21649561211047804. eCollection 2021. PMID 34917419
- [Result] Park ER, Perez GK, Millstein RA, Luberto CM, Traeger L, Proszynski J, Chad-Friedman E, Kuhlthau KA. A Virtual Resiliency Intervention Promoting Resiliency for Parents of Children with Learning and Attentional Disabilities: A Randomized Pilot Trial. Matern Child Health J. 2020 Jan;24(1):39-53. doi: 10.1007/s10995-019-02815-3. PMID 31650412

DOCUMENTS (2):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT05535348/Prot_000.pdf
  • Informed Consent Form (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT05535348/ICF_001.pdf